CLINICAL TRIAL: NCT01348776
Title: The Efficiency of the Hair2Go Device: A Prospective, Open, Label Study With Before-After Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Syneron Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHR-2
Record Dates: First submitted 2011-05-02; First posted 2011-05-05 (Estimated); Results first posted 2013-04-04 (Estimated); Last update posted 2013-04-04 (Estimated); Status verified 2013-04

CONDITIONS: Hair Removal
Keywords: hair reduction; hair removal; hair clearance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hair2Go (Mē) (Experimental): Subjects treated with Hair2Go (Mē) Device
  Interventions: Device: Hair2Go (Mē)

INTERVENTIONS:
Device: Hair2Go (Mē) — Treatment with Hair2Go Device 7 times every week with maintenance treatments once a month for 3 months
  Other Names: Mē my elōs

SUMMARY:
The purpose of this study is to determine efficiency of Hair2Go device for short-term and long-term removal of unwanted hair adjunctive to shaving using a before-after study design.

DETAILED DESCRIPTION:
This study is a multicenter study, designed to determine the efficacy of the Hair2Go hair removal device and to compare the extent of hair removal with and without maintenance treatments. Preferably, two anatomical regions to be treated will be selected including the axilla and either the legs (calves) or forearms. The size of the area treated will be approximately 5x5 cm2. Additional areas including the face can be treated according to the subject's request with the PI's discretion but are not mandatory. Subjects will be provided with the device and will be instructed as to the method of usage. The subjects will be expected to self-administer the treatment at the clinic in a "simulated home environment". The duration of the treatment session is approximately 30-60 minutes. Each of the selected anatomical regions (both left and right sides) will be treated with either low, medium, or high Elōs energy level according to the PI's discretion. However all anatomical regions except for the axilla will be treated with either low or medium elōs energy levels only. Only the axilla will be treated up to an energy of 4J//cm2 A defined area of 5x5 cm2cm2 in the leg will not be treated and will serve as a reference for the temporal changes in hair growth that might be subject to factors, including fluctuations in hormone levels. Both sides (left and right) of the same anatomical region will receive the basic treatments. One side will receive 3 additional maintenance treatments in 4 week intervals ("Maintenance" vs "No maintenance" side) until the end of the experiment. More specifically, the study includes up to 11 visits at the clinic: initial consultation, 7 basic treatments in 1 week intervals followed in one side by 3 maintenance treatments, each 4 weeks apart. Follow ups will be conducted at 4 and 12 weeks after the last basic treatment.

ELIGIBILITY:
Inclusion Criteria

1. Healthy males and females, between 18 and 65 years of age.
2. Subject has Black or dark brown terminal hairs in the areas to be treated.
3. Terminal hair density requirement of greater than 15 hairs within the hair count site (3x3 cm area) as determined by manual hair count performed by the study investigator.
4. Willing to sign informed consent.
5. Willing to follow the treatment schedule and post treatment follow-up.
6. Willingness to have photographs of the treated area taken that may be used for marketing and educational presentation and/or publications
7. Willingness to avoid excessive sun exposure two weeks prior to treatments

Exclusion Criteria

Skin and Hair

1. Subjects with white, red, light brown and/ or blonde hairs in the areas to be treated.
2. A history of keloidal scarring (hypertrophic scars or keloids).
3. Active dermatologic lesion or infection in the treatment site.
4. Subject has permanent tattoos or makeup in the treatment area.
5. Recently tanned in the area to be treated and/or unable or unlikely to refrain from tanning during the study.
6. Subject has disease related to photosensitivity, such as porphyria, polymorphic light eruption, solar urticaria, lupus, etc
7. Subject has a history of herpes outbreak in the area of treatment, unless receiving preventative treatment from physician

   Other Medical Conditions
8. Pregnant, planning to become pregnant, hormone fluctuations and/or breast feeding during the experiment.
9. Subjects with Diabetes (Type I or II) or other systemic or metabolic condition
10. Subject has an active electrical implant anywhere in the body, such as a pacemaker, an internal defibrillator, insulin pump, incontinence device, etc.
11. Subject suffers from epilepsy.
12. Subject has active cancer, or has a history of skin cancer or any other cancer in the area to be treated, including presence of malignant or pre-malignant pigmented lesions.
13. Subject received radiation therapy or chemotherapy treatments with the past 3 months.
14. Subject has known anticoagulative or thromboembolic condition or is on any form of anticoagulation treatment.
15. Subject has a history of immunosuppressant/immune deficiency disorders (including HIV infection or AIDS) or currently using immunosuppressive medications.
16. Subject has any other condition which in the physician's opinion would make it unsafe for the subject to be treated.

    Medication/treatments
17. Subject had rotating type tweezer epilator treatment, or waxing within the last 3 weeks
18. Subject had electrolysis treatment within the last 6 months over the treatment area.
19. Subject had any type of professional intense pulsed light (IPL), laser or RF hair removal in the treatment site within the last 6 months.
20. Subject is taking medication known to induce photosensitivity, including non-steroidal anti-inflammatory agents, tetracyclines, phenothiazines, thiazide diuretics, sulfonylureas, sulfonamides, Dacarbazine(DTIC), fluorouracil, vinblastine, and griseofulvin within 4 weeks of therapy.
21. Subject has been taking Accutane® within 6 months of therapy.
22. Subject has been on steroid regimen during the last three months.
23. Subject is on Gold therapy (for arthritis treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2011-03; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerome M Garden, MD, Principal Investigator — Northwestern Memorial Hospital; Vince Afsahi, MD, Principal Investigator — South Coast Dermatology Institute; Brian D Zelickson, MD, Principal Investigator — Abbot Northwestern Hospital Center for Cosmetic Care; Michael Gold, MD, Principal Investigator — Tennessee Clinical Research Center
Locations (4):
- United States (4):
  - South Coast Dermatology, Tustin, California
  - Dr Jerome Garden, Chicago, Illinois
  - Zel Skin and Laser Specialist, Edina, Minnesota
  - Tennessee Clinical Research Center, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment was conducted in a medical clinic. The recruitment continued from April to October 2011.
Pre-assignment Details: 3 subjects were found not eligible and 1 withdrew the informed consent before beginning treatments.
Groups:
- Hair2Go (Me): Subjects treated with the Hair2Go (Me) Device
Period: Overall Study
Arm/Group | Hair2Go (Me)
Started | 87 (3 subjects were lost to follow-up: 2 after the 1-month follow-up, 1 after performing 4 treatments)
Completed | 84
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Hair2Go (Me)
Number analyzed (Participants) | 87
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 87
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.4 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79
  Male | 8
Region of Enrollment [Number; unit: participants]
  United States | 87

OUTCOME MEASURES:

1. Primary Outcome: Hair Clearance 1 Month After Last Treatment
Description: Hair clearance = the percent of hair cleared from baseline to endpoint.
Time Frame: 3 months (1 month after 7 weekly treatments)
Population: Sample size was discussed with the FDA during a pre-IDE meeting.
Measure: Mean (Standard Deviation); unit: %baseline hair count
Units Other Than Participants: areas of treatment
Groups:
- Hair2Go (Mē) Maintenance Side (Before Maintenance Tx): Subjects treated with Hair2Go (Mē) Device:the treatment areas include the side that is randomized to receive maintenance treatments. This time point is before maintenance treatments were given.
- Hair2Go (Mē) no Maintenance Side: Subjects treated with Hair2Go (Mē) Device:the treatment areas include the side that is randomized NOT to receive maintenance treatments.
Arm/Group | Hair2Go (Mē) Maintenance Side (Before Maintenance Tx) | Hair2Go (Mē) no Maintenance Side
Number analyzed (Participants) | 87 | 87
Number analyzed (areas of treatment) | 143 | 143
%baseline hair count | 56.83 (42.96) | 54.08 (41.21)

2. Secondary Outcome: Hair Clearance at 3-month (Final) Follow up
Description: Hair clearance = %hair cleared from baseline to endpoint after 7 weekly treatments with or without additional 2 monthly maintenance treatments.
Time Frame: 5 months (3 months after 7 weekly treatments)
Population: All areas with photos that allowed reliable hair counting were included for this analysis.
Measure: Mean (Standard Error); unit: %baseline hair count
Units Other Than Participants: Treatment Areas
Groups:
- Maintenance Side: Hair clearance after 7 weekly treatments+2 additional monthly maintenance treatments
- No Maintenance Side: Hair clearance after 7 weekly treatments without additional maintenance treatments
Arm/Group | Maintenance Side | No Maintenance Side
Number analyzed (Participants) | 87 | 87
Number analyzed (Treatment Areas) | 142 | 139
%baseline hair count | 58.3 (37.4) | 44.2 (38.4)

3. Secondary Outcome: Occurrence of Anticipated Effects on Skin
Description: As with other IPL devices, subjects were informed that they should expect some sense of warmth, tingling, or itching, when the device was applied. This was anticipated to be mild to moderate. Subjects could also expect transient erythema and edema at the treatment site that usually disappears within 24 hours.
Time Frame: Up to 19 weeks
Measure: Number; unit: Number of reports
Units Other Than Participants: total treatments
Groups:
- Anticipated Skin Effects: Anticipated skin effects included mild to moderate sense of warmth, tingling, or itching, and transient erythema and edema.
Arm/Group | Anticipated Skin Effects
Number analyzed (Participants) | 87
Number analyzed (total treatments) | 2765
Number of reports
  Erythema | 20
  Pruritis | 2
  Edema | 2
  Inflammation | 2

4. Secondary Outcome: Tolerability Level of the Procedure Following Treatments
Description: Gathering information about the tolerability of the procedure following weekly treatments 1, 3, 7 and maintenance treatment 3 by asking subjects to rate the tolerability of the procedure based on 5 point pain scale (no pain, mild pain, moderate pain, severe pain, Intolerable [had to stop treatment]) .
  The distribution of the tolerability level is based on the analysis of the areas treated and not on the number of participants since each participant was treated on more than one area. Therefore the number of treated areas exceeds the number of participants and the unit of measurement is % treated areas that were rated.
Time Frame: 1, 3, 7 weeks (basic weekly treatment 1, 3, and 7), and 5 months (maintenance monthly treatment#3)
Measure: Number; unit: % treated areas
Units Other Than Participants: Treatment areas analyzed
Groups:
- Treatment #1: Self assessment of tolerability level of procedure during 1st treatment
- Treatment #3: Self assessment of tolerability level of procedure during 3rd treatment
- Treatment #7: Self assessment of tolerability level of procedure during 7th treatment
- Maintenance Treatment #3: Self assessment of tolerability level of procedure during 3rd maintenance treatment
Arm/Group | Treatment #1 | Treatment #3 | Treatment #7 | Maintenance Treatment #3
Number analyzed (Participants) | 87 | 87 | 87 | 87
Number analyzed (Treatment areas analyzed) | 332 | 330 | 330 | 146
% treated areas
  No Pain | 83.13 | 91.52 | 89.09 | 86.99
  Mild Pain | 13.86 | 8.48 | 8.48 | 11.64
  Moderate Pain | 3.01 | 0 | 2.42 | 1.37
  Severe Pain | 0 | 0 | 0 | 0
  Intolerable (had to stop treatment) | 0 | 0 | 0 | 0

5. Secondary Outcome: Subject Satisfaction
Description: Gathering information about the subject satisfaction from the hair removal procedure based on 5 point satisfaction scale.
Time Frame: 5 months (final follow up)
Population: Two subjects did not report on satisfaction.
Measure: Number; unit: participants
Groups:
- Hair2Go (Mē): Subjects treated with the Hair2Go (Me) Device
Arm/Group | Hair2Go (Mē)
Number analyzed (Participants) | 85
participants
  Very satisfied | 31
  Satisfied | 33
  Slightly satisfied | 9
  No opinion | 4
  Unsatisfied | 8

ADVERSE EVENTS:
Time Frame: 5 month - from 1st treatment to last follow up
Arm/Group | Hair2Go (Me)
Serious Adverse Events (participants affected / at risk) | 0/87
Other Adverse Events (participants affected / at risk) | 3/87
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hair2Go (Me) (N=87)
Blister (Skin and subcutaneous tissue disorders) | 1 (2)
Severe Pain (Skin and subcutaneous tissue disorders) | 2 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days